CLINICAL TRIAL: NCT02033733
Title: Post-arrest Therapeutic Hypothermia. Does Use of Neuromuscular Blockers Achieve Faster Cooling Time?
Brief Title: When Cooling a Patient After Cardiac Arrest, Does Use of a Neuromuscular Blocking Agent Make Your Job Easier?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Eyad AlThenayan, Dr. Eyad AlThenayan, University of Western Ontario, Canada
Other Study IDs: 5511
Record Dates: First submitted 2014-01-04; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Postcardiac Arrest Therapeutic Hypothermia
Keywords: Post cardiac arrest; Postcardiac arrest therapeutic hypothermia; Therapeutic hypothermia protocol; Neuromuscular blocking agents; Muscle relaxants; Hypothermia-induced increased muscle tone; Microshivering
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adequate cooling time: Patients that reached target temperature within 4 hours of initiation of the hypothermia protocol will be in the "adequate cooling time" group.
  Interventions: Drug: Cisatracurium infusion; Drug: Cisatracurium prn bolus
- Inadequate cooling time: Patients that did not reach target temperature within 4 hours of initiation of the hypothermia protocol will be in the "inadequate cooling time" group.
  Interventions: Drug: Cisatracurium infusion; Drug: Cisatracurium prn bolus

INTERVENTIONS:
Drug: Cisatracurium infusion — This group will include postcardiac arrest patients that have received a cisatracurium infusion as part of their therapeutic hypothermia protocol. It will only include patients that had their infusion started within 2 hours from protocol initiation. Patients that received an infusion as a rescue measure (beyond the first 2 hours) or did not receive and infusion at all will not be included in this group.
  Most patients admitted to our ICU postcardiac arrest prior to October 2011, will likely belong to this group (the cisatracurium infusion group).
  Other Names: Neuromuscular blocking agent infusion; NMBA infusion; Continuous NMBA infusion; Continuous cisatracurium infusion; Cisatracurium by continuous infusion
Drug: Cisatracurium prn bolus — Patients that have not received a cisatracurium infusion within the first 2 hours from protocol initiation will be in this group. These are likely to be patients admitted to our ICU after October 2011 (when the protocol change happened).
  Other Names: neuromuscular blocking agent prn bolus; NMBA prn bolus; cisatracurium intermittent bolus; intermittent bolus administration of cisatracurium

SUMMARY:
After successful resuscitation from cardiac arrest, cooling the whole body is a well established treatment that improves the chances of the brain recovering. This however, has to be done within a certain time-frame from the arrest. The purpose of this study is to explore the best way of dosing the muscle relaxing medications that are given during the cooling process.

Hypothesis: In the context of our institutional therapeutic hypothermia protocol, cisatracurium infusions lead to faster drops in core temperature when compared to cisatracurium prn boluses alone.

DETAILED DESCRIPTION:
STUDY RATIONALE:

A large proportion of comatose survivors of cardiac arrest presenting to our intensive care units at London Health Sciences Centre (LHSC) undergo therapeutic hypothermia. Current evidence suggests that timely achievement of target temperatures is desirable to improve outcomes. At LHSC, this intervention is protocolized with a defined set of preprinted orders that includes a dosing regimen for neuromuscular blocking agents (NMBA's). Our preprinted protocol has been in place since January of 2004. Cisatracurium infusions were part of the therapeutic hypothermia protocol until October 2011. Since that time, our protocol has changed to cisatracurium prn boluses for any observed shivering. In this study we will examine if there has been any change in the times to achieving target temperatures with the implementation of this change. It is important to note that no other change in our protocol has taken place since it was first implemented, making our before and after comparison valid and fair.

Our hypothesis is that NMBA infusions lead to a faster drop in core temperatures when compared to NMBA prn boluses. If this were to stand true, we would expect cisatracurium IV infusions to result in faster reductions in core temperature when compared with cisatracurium prn boluses in the context of our therapeutic hypothermia protocol. Hypothermia has been known to cause a subclinical increase in muscle tone. This previously reported phenomenon has been named "microshivering". When attempting to reduce core temperatures, microshivering is likely a natural body response to try to restore body temperature back to normal. We therefore hypothesize that NMBA infusions are likely more effective at abolishing microshivering, which would be a desirable effect when trying to induce therapeutic hypothermia.

Although current American Heart Association (AHA) guidelines suggest considering the administration of NMBA's to facilitate induced hypothermia and control shivering. Their recommendation is to minimize the duration of NMBA use or if possible, avoid them altogether. After the publication of these guidelines our institutional protocol changed to prn boluses instead of the previous infusion orders. We therefore believe it is important to examine the effects of this change on our cooling protocol and potentially add to the growing body of knowledge in this field.

ELIGIBILITY:
Inclusion Criteria:

* Admission to adult ICU (age ≥18 years) at London Health Sciences Centre
* Primary reason for ICU admission: postcardiac arrest
* Both in-hospital and out-of-hospital cardiac arrest will be included
* ICU admission between Jan 2008 and Dec 2012.

Exclusion Criteria:

- ICU admissions primarily for reasons other than cardiac arrest.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the intensive care unit (ICU) with a diagnosis of postcardiac arrest between Jan 2008 and Dec 2012 will be examined.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Time to attaining target temperature (hours). | From initiation of hypothermia protocol to reaching a core body temperature of ≤34ºC, assessed up to 72 hours from protocol initiation.
  The primary outcome will be a binary outcome that is: adequate cooling time versus inadequate cooling time based on the time needed to achieve target temperatures. We will define adequate cooling time as being ≤ 4 hours from initiation of protocol to reaching target temperature. Inadequate cooling time will be requiring > 4 hours to achieve that goal. Target core body temperature range in our institutional protocol is 32 - 34ºC.
  The primary outcome will be assessed using a logistic regression model, constructed using covariates affecting speed of cooling as determined by expert opinion and current evidence apriori. The variables will be age, sex, weight, pre-protocol core body temperature, initial arrest rhythm and infusion versus boluses. The model will be used to determine whether the cisatracurium dosing regimen is an independent predictor of adequate patient cooling time or not.

SECONDARY OUTCOMES:
Cerebral performance category score on hospital discharge. | Upon discharge from hospital, assessed up to 36 months postcardiac arrest.
  Neurological outcome on discharge from hospital as defined by the cerebral performance category (CPC) scale. The CPC scale is a 5 point scale. The outcome measure will be dichotomized into good or bad. Good outcome will be equivalent to CPC scores of 1 & 2 (where the patient is independent), and bad outcome will be equivalent to CPC scores of 3, 4 & 5 (where the patient is either dependent or dead). We will examine whether the use of a neuromuscular blocking agent infusion correlates with good CPC scores on hospital discharge or not.
  CPC Scale:
  1. Functioning normally and independent, possibly with a minor disability.
  2. Moderately disabled, still independent.
  3. Conscious but with a severe disability, dependent.
  4. Unconscious (comatose or in a persistent vegetative state).
  5. Brain dead or dead by traditional criteria.
Hospital length of stay postcardiac arrest (days). | Days spent in hospital after successful resuscitation from cardiac arrest, assessed up to 36 months from the date of cardiac arrest
  Hospital length of stay (LOS) post-cardiac arrest will be calculated from the day of the cardiac arrest to the day of hospital discharge. If prior to the arrest the patient was an inpatient, we will only count the days from the arrest to discharge. Days spent in hospital prior to the arrest will not be included.
Intensive care unit length of stay postcardiac arrest (days). | Days spent in the intensive care unit after successful resuscitation from cardiac arrest, assessed up to 36 months from the date of cardiac arrest.
  The length of stay (LOS) in the intensive care unit (ICU) after successful resuscitation from cardiac arrest in days.

OTHER OUTCOMES:
Time required to normalize lactate (hours) | Time from a sustained return of spontaneous circulation to the first recorded normal lactate level, assessed up to 7 days (168 hours) postcardiac arrest.
  Neuromuscular blocking agent (NMBA) infusions are likely to abolish microshivering and hence reduce lactate generation. This is likely to reduce the times needed for patients to normalize their lactate levels post resuscitation from cardiac arrest. We will examine whether NMBA infusions were associated with better lactate clearance rates (shorter times to normalization of lactate levels) in comparison to NMBA prn boluses or not.

CONTACTS AND LOCATIONS:
Overall Officials: Eyad Althenayan, MD, Principal Investigator — Western University, Canada; Philip Jones, MD, FRCPC, Study Director — Western University, Canada; Bryan Young, MD, FRCPC, Study Chair — Western University, Canada; Ahmed F Hegazy, MD, FRCPC, Study Director — Western University, Canada; Ana Igric, MD, FRCSC, Study Director — Western University, Canada; Carolyn Benson, MD, Study Director — Western University, Canada
Locations (2):
- Canada (2):
  - University Hospital, London Health Sciences Centre, University of Western Ontario, London, Ontario
  - Victoria Hospital, London Health Sciences Centre, University of Western Ontario, London, Ontario

REFERENCES:
- [Background] Sendelbach S, Hearst MO, Johnson PJ, Unger BT, Mooney MR. Effects of variation in temperature management on cerebral performance category scores in patients who received therapeutic hypothermia post cardiac arrest. Resuscitation. 2012 Jul;83(7):829-34. doi: 10.1016/j.resuscitation.2011.12.026. Epub 2012 Jan 8. PMID 22230942
- [Background] Werlhof V, Sessler DI. Pancuronium does not decrease oxygen consumption during hypothermic or normothermic cardiopulmonary bypass. Anesth Analg. 1995 Sep;81(3):465-8. doi: 10.1097/00000539-199509000-00006. PMID 7653805
- [Background] Peberdy MA, Callaway CW, Neumar RW, Geocadin RG, Zimmerman JL, Donnino M, Gabrielli A, Silvers SM, Zaritsky AL, Merchant R, Vanden Hoek TL, Kronick SL; American Heart Association. Part 9: post-cardiac arrest care: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S768-86. doi: 10.1161/CIRCULATIONAHA.110.971002. PMID 20956225